CLINICAL TRIAL: NCT06262165
Title: BILAN: Evaluation of Liver Damage in Patients With Anorexia Nervosa by Blood BIomarker ANaLysis
Brief Title: Evaluation of Liver Damage in Patients With Anorexia Nervosa by Blood Biomarker Analysis
Acronym: BILAN
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC23_0497
Record Dates: First submitted 2024-01-29; First posted 2024-02-15 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-01

CONDITIONS: Anorexia Nervosa
Keywords: Biomarkers; Liver fibrosis; Liver steatosis; Anorexia nervosa; Enteral refeeding
MeSH Terms: conditions — Anorexia Nervosa; Liver Cirrhosis; Fatty Liver

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients with Anorexia Nervosa — Patients with Anorexia Nervosa hospitalized for malnutrition

SUMMARY:
The main goal of the BIocoLlection in Anorexia Nervosa-liver damage evaluation BILAN study the blood biomarkers associated with liver cytolysis.

DETAILED DESCRIPTION:
Study of the association between blood biomarkers and the presence of hepatic cytolysis, defined by AST and/or ALT above normal.

ELIGIBILITY:
Inclusion Criteria :

* Patient over 15 years old
* Diagnosis of Restricted Eating Disorders including Anorexia Nervosa according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
* Admission to Nantes University Hospital.

Exclusion Criteria :

* Chronic active viral hepatitis
* Hemochromatosis
* Other genetic, autoimmune.
* Treatment with a drug known to induce fatty liver disease (amiodarone, carbamazepine, tamoxifen, valproate, clozapine, anti-retrovirals) unless the dose has been stable for ≥ 3 months
* Excessive alcohol consumption (≥ 30 grams per day in men, ≥ 20 grams per day in women)
* Pregnant, parturient or breast-feeding women, persons deprived of liberty, adults under legal protection or unable to express their consent, persons not affiliated or not beneficiaries of a social security scheme, persons under guardianship or curators

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive inclusion of patients hospitalized in the endocrinology department for anorexia nervosa with malnutrition criteria.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2032-06-15 (Estimated); Study Completion 2032-12-15 (Estimated)

PRIMARY OUTCOMES:
Identification of new blood biomarkers and hepatic cytolysis | Two years
  Identify changes in concentration of new blood biomarkers in patients suffering from hepatic cytolysis, defined by aspartate transaminases (AST) and/or alanine transaminases (ALT) above normal values, compared to those with normal enzyme levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided